CLINICAL TRIAL: NCT01292213
Title: Identification and Characterisation of Bacteria Causing Chronic Cough Among Children in the United Kingdom
Brief Title: A Study to Identify and Characterise Bacteria Causing Chronic Cough Among Children in United Kingdom
Status: Terminated | Type: Observational
Why Stopped: • Long delay due to challenges with sample analysis at local labs; • Low recruitment of case and control subjects; • Constant staff turn-over in the sites.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112956
Record Dates: First submitted 2011-02-03; First posted 2011-02-09 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Infections, Respiratory Tract
Keywords: Chronic cough; Haemophilus influenzae
MeSH Terms: conditions — Respiratory Tract Infections; Chronic Cough; Haemophilus Infections | interventions — Blood Specimen Collection; Bronchoscopy; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cough swab, oropharyngeal swab, nasopharyngeal swabs, blood and bronchoscopy/ bronchoalveolar lavage samples.

GROUPS / COHORTS (2):
- Cases: Subjects diagnosed with chronic cough who are undergoing general anaesthesia and bronchoscopy/BAL as part of the diagnostic process for chronic cough.
  Interventions: Procedure: Cough swab; Procedure: Oropharyngeal swab; Procedure: Nasopharyngeal swabs; Procedure: Blood sample; Procedure: Bronchoscopy/ bronchoalveolar lavage samples; Other: Data collection
- Controls: Subjects without respiratory symptoms who are undergoing general anaesthesia for elective surgery or endoscopy of non-respiratory-related conditions.
  Interventions: Procedure: Cough swab; Procedure: Oropharyngeal swab; Procedure: Nasopharyngeal swabs; Procedure: Blood sample; Procedure: Bronchoscopy/ bronchoalveolar lavage samples; Other: Data collection

INTERVENTIONS:
Procedure: Cough swab — Samples will be tested to determine and characterise the bacteria that may be associated with chronic cough.
Procedure: Oropharyngeal swab — Samples will be tested to determine and characterise the bacteria that may be associated with chronic cough.
Procedure: Nasopharyngeal swabs — Samples will be tested to determine and characterise the bacteria and viruses that may be associated with chronic cough.
Procedure: Blood sample — Samples will be tested to determine and characterise the immunological markers that may be associated with chronic cough.
Procedure: Bronchoscopy/ bronchoalveolar lavage samples — Samples will be tested to determine and characterise the bacteria, viruses and immunological markers that may be associated with chronic cough.
Other: Data collection — Questionnaire completion.

SUMMARY:
The purpose of this study is to investigate the role of Haemophilus influenzae and other bacteria in causing chronic cough, through a direct comparison of chronic cough cases and healthy controls recruited from paediatric respiratory clinics in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/ legally acceptable representative can and will comply with the requirements of the protocol.
* A male or female child between, and including, six to 72 months of age at the time of enrolment.
* Written informed consent obtained from the parent(s)/ legally acceptable representative of the subject.
* No antibiotic therapy within four weeks prior to the visit.
* No cystic fibrosis or known major immunodeficiency such as agammaglobulinaemia, T cell deficiency or Human Immunodeficiency Virus / Acquired Immune Deficiency Syndrome.
* No documented evidence or suspicion of gastroesophageal reflux disease.
* No evidence of an upper viral respiratory infection four weeks prior to the visit.

In addition, all subjects regarded as 'cases' must satisfy all the following criteria at study entry:

* Persistent cough greater than eight weeks.
* No response to five-day prednisolone treatment.
* Chest X-ray showing no evidence of a lobar pneumonia or gross structural abnormality.

In addition, all subjects regarded as 'controls' must satisfy the following criteria at study entry:

* No respiratory symptoms four weeks prior to the visit.
* No documented evidence or suspicion of lung disease upon physical examination.

Exclusion Criteria:

* Concurrently participating in another study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Use of any investigational or non-registered product within 30 days prior to study procedures, or planned use during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Child in care.

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged six to 72 months, residing in the United Kingdom. These children will be classified as cases and controls.
  Cases will be children who have had persistent cough for greater than eight weeks and are undergoing general anaesthesia for clinically indicated bronchoscopy/ bronchoalveolar lavage as part of the diagnostic process for chronic cough.
  Controls will be children who are undergoing general anaesthesia with endotracheal intubation for elective surgery or endoscopy for non-respiratory-related conditions and had no acute or chronic respiratory symptoms during the four weeks prior to the visit.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of Haemophilus influenzae, in the absence of co-infection with other bacteria, in the lower airways of cases and controls | 12-15 months from study initiation

SECONDARY OUTCOMES:
Occurrence of Haemophilus influenzae, regardless of co-infection with other bacteria, in the lower airways of cases and controls | 12-15 months from study initiation
Occurrence of Streptococcus pneumoniae in the lower airways of cases and controls | 12-15 months from study initiation
Occurrence of Haemophilus influenzae in cough swabs and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Occurrence of Haemophilus influenzae in the lower airways and/or nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Bacterial load of Haemophilus influenzae in the lower airways and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Occurrence of Haemophilus haemolyticus in the lower airways and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Antimicrobial resistance of Haemophilus influenzae in lower airways | 12-15 months from study initiation
Occurrence of viral pathogens in the lower airways and nasopharynx of cases and controls | 12-15 months from study initiation
Occurrence of Moraxella catarrhalis in the lower airways of cases and controls | 12-15 months from study initiation
Occurrence of other bacterial pathogens in the lower airways of cases and controls | 12-15 months from study initiation
Occurrence of Streptococcus pneumoniae in cough swabs and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Occurrence of Moraxella catarrhalis in cough swabs and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Occurrence of Streptococcus pneumoniae in the lower airways and/or nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Occurrence of other bacterial pathogens in the lower airways and/or nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Bacterial load of Streptococcus pneumoniae in the lower airways and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Bacterial load of Moraxella catarrhalis in the lower airways and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Occurrence of serotypes of Haemophilus influenzae in the lower airways and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Occurrence of serotypes of Streptococcus pneumoniae in the lower airways and nasopharynx/ oropharynx of cases and controls | 12-15 months from study initiation
Antimicrobial resistance of Streptococcus pneumoniae in lower airways | 12-15 months from study initiation
Antimicrobial resistance of Moraxella catarrhalis in lower airways | 12-15 months from study initiation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Sheffield